CLINICAL TRIAL: NCT05517850
Title: Comprehensive Therapist-guided Cognitive Behavioral Therapy for Atopic Dermatitis Versus a Shortened Digital Self-care Intervention: A Randomized Non-Inferiority Trial
Brief Title: Therapist-guided vs Self-guided CBT for AD: Non-inferiority Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Martin Kraepelien, Licensed clinical psychologist, Principal investigator, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBTADNI
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
Keywords: Cognitive behavioral therapy; Self-guided intervention; Digital intervention; Exposure therapy
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will know about the randomization to one of two types of cognitive behavioral therapy. Participants will have no way to know their assignment beforehand, or the defining characteristics of either condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapist-guided (Active Comparator): 12 weeks of therapist-guided, exposure-based intervention via tha internet, with comprehensive material
  Interventions: Behavioral: Therapist-guided cognitive behavioral therapy administered online
- Self-guided (Experimental): 12 weeks of self-guided, exposure-based intervention via the internet, with shortened and improved material
  Interventions: Behavioral: Self-guided digital intervention based on cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Therapist-guided cognitive behavioral therapy administered online — This intervention consists of 10 modules of education and interventions and lasts 12 weeks. An introduction provides information about CBT and AD. Step by step, the participants are introduced to the proposed active treatment components: mindfulness training, and exposure with response prevention. Through this whole process, the participant is guided by a therapist. The therapist may be contacted through a secure internet platform at any time and responds within 48 hours. Participants reads the education material, construct exercises to perform, describes their progress in homework assignments, and receives feedback from their therapist.
  Arms: Therapist-guided
Behavioral: Self-guided digital intervention based on cognitive behavioral therapy — Participants will access a digital platform, read information, and perform exercises in their everyday life. The main treatment components are mindfulness and exposure with response prevention, with a specific focus on itch. Participants will be able to practice mindfulness with the help of instructions and examples. Participants will receive detailed instructions and guidance, and get to choose exposure exercises from a long list of examples. Participants will also be free to create their own relevant exposure situations within the intervention. Digital self-care consists of 8 modules. The only active interventions, mindfulness and exposure are introduced week 1 and 2, respectively. From week 3-7, no new interventions are introduced and participants are advised to continue practicing the interventions, but there is a new theme of education each week, to act as inspiration for exercises. The last 4 weeks, the participant is merely advised to continue practice.
  Arms: Self-guided

SUMMARY:
The study aims to test the hypothesized non-inferiority of a self-guided digital intervention compared to a therapist-guided variant for people with atopic dermatitis (AD). Both interventions are based on Cognitive behavioral therapy. Participants will be recruited from advertisements in social media. Measurements of AD symptoms and psychological well-being will be conducted at pre-treatment, post-treatment as well as 6-month and one-year follow-up.

DETAILED DESCRIPTION:
Background: Digital self-care based on Cognitive-behavioral therapy (CBT) could be an effective alternative to guided CBT for people with atopic dermatitis (AD) and has the theoretical potential to significantly increase access to psychological treatment for patients with AD, whilst being cost-effective for health care organizations.

Aim: To investigate whether a shortened digital self-care intervention is noninferior to, and cost-effective compared with, a comprehensive and therapist-guided CBT treatment for AD.

Intervention: Participants randomized to guided care will receive internet-delivered cognitive behavior therapy for 12 weeks. Participants randomized to digital self-care will have access to a self-guided intervention for 12 weeks_

Design, setting, and participants: This is a single-blind, randomized clinical non-inferiority trial at Karolinska Institutet, a medical university in Stockholm, Sweden. 174 adult participants with AD will be recruited through self-referral. Participants will be randomized 1:1 to the two experimental conditions. At post-treatment (primary endpoint), non-inferiority will be tested and resource use will be compared between the two treatment groups. Cost-effectiveness will be explored at 1-year follow-up. Potential mediators will be investigated. Data will be analyzed intention-to-treat.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported AD diagnosed by physician (potential participants will disclose the circumstances of their diagnosis)
* No new types of medications introduced for six months prior, with no intention of future change
* Able to understand Swedish
* Access to the internet and a smartphone

Exclusion Criteria:

* Other disease or condition that has immediate treatment priority over AD. This could be an ongoing demanding treatment of a severe somatic or psychiatric condition. No specific diagnoses are inevitably a cause for exclusion, as potential participants will rather be evaluated on a case-to-case basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in atopic dermatitis symptoms | Change from pre-treatment (baseline) to post-treatment (week 12); weekly (week1-11); change from pre-treatment (baseline) to 6 month follow-up (week 36); change from pre-treatment (baseline) to 1 year follow-up (week 60)
  Patient oriented eczema scale (POEM). 7 items. Higher scores indicate greater severity of eczemic symptoms. Scores range from 0 to 28.

SECONDARY OUTCOMES:
Change in itching sensation | Change from pre-treatment (baseline) to post-treatment (week 12); weekly (week1-11); change from pre-treatment (baseline) to 6 month follow-up (week 36); change from pre-treatment (baseline) to 1 year follow-up (week 60)
  Peak pruritus rating scale (NRS). 2 items. Higher scores indicate more severe itch. Scores range from 1-10
Change in stress reactivity | Change from pre-treatment (baseline) to post-treatment (week 12); weekly (week1-11); change from pre-treatment (baseline) to 6 month follow-up (week 36); change from pre-treatment (baseline) to 1 year follow-up (week 60)
  Perceived stress scale (PSS). 14 items. Higher scores indicate more stressed mood and greater reactivity. Score ranges from 0-56.
Change in depressive symptoms | Change from pre-treatment (baseline) to post-treatment (week 12); weekly (week1-11); change from pre-treatment (baseline) to 6 month follow-up (week 36); change from pre-treatment (baseline) to 1 year follow-up (week 60)
  Patient Health Questionnaire.(PHQ-9). 9 items. Higher total scores indicate greater severity of depression. Scores range from 0 to 27.
Change in skin-related quality of life | Change from pre-treatment (baseline) to post-treatment (week 12); weekly (week1-11); change from pre-treatment (baseline) to 6 month follow-up (week 36); change from pre-treatment (baseline) to 1 year follow-up (week 60)
  Dermatological Life Quality Index (DLQI). 10 items. Higher score indicate lower quality of life related to skin symptoms.Scores range from 0 to 30.
Change in insomnia symptoms | Change from pre-treatment (baseline) to post-treatment (week 12); weekly (week1-11); change from pre-treatment (baseline) to 6 month follow-up (week 36); change from pre-treatment (baseline) to 1 year follow-up (week 60)
  Insomnia severity index (ISI). 7 items. Higher scores indicates more severe insomnia. Scores range from 0 to 28.
Treatment credibility | 2 weeks after treatment start (baseline).
  Credibility/expectancy questionnaire (CEQ). The CEQ ranges from 0 to 10 points per item and 0 to 50 points in total, where a higher score reflects better treatment credibility.
Intervention satisfaction | Post-treatment (12 weeks)
  Client Satisfaction Questionnaire (CSQ-8). Scores range from 8-32 with higher scores indicating greater satisfaction. An average Client Satisfaction Questionnaire-8 score of at least 22 will provide support for the acceptability and feasibility of this intervention.
Quality of life for health economy analysis | Post treatment (week 12) to one-year follow-up (week 60)
  Euro quality of life 5 dimensions (EQ5D). 5 items. Higher scored indicate higher quality of life. A calculation gives a total score from 0 to 100.
Health economics | Change from pre-treatment (baseline) to post-treatment (week 12); change from pre-treatment (baseline) to 6 month follow-up (week 36); change from pre-treatment (baseline) to 1 year follow-up (week 60)
  Treatment Inventory of Costs in Psychiatric Patients (TIC-P)
Post-treatment adherence to exposure exercises | Post-treatment (12 weeks)
  Time spent on exercises (ToE) Adherence to the exposure exercises will be determined by an online questionnaire where it will be stated on a four point Likert scale will state to what extent participants have worked with exposure: "not at all", "occasionally", "more than half of the days" and "daily". Acceptable level of adherence will be set to at least 50 % of participants working actively with exposure a majority of the days during a week for 4 weeks or more.
Usability | Post-treatment (12 weeks)
  The System Usability Scale (SUS). The SUS consists of ten items, with a range of 0-4 points per item. The items are summed up and calculated with a formula resulting in a total score between 0 and 100, with a higher score reflecting better system usability.
Adverse events | Post-treatment (12 weeks)
  Adverse events (AE). Participants are asked if they have had an adverse event as a result of treatment, and if so to describe it. If they have experienced more than oneadverse event, the question is repeated.
Time spent on treating | From week 1 to 12, throughout
  Time spent on treatment (ToT): Time in minutes spent by therapists on writing messeges, phone calls, etc.

OTHER OUTCOMES:
Telephone interview | Post treatment (12 weeks)
  A semi-structured interview concerning the experience of the intervention and format will be conducted via telephone

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for psychatry research, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual data will be available upon reasonable request.

REFERENCES:
- [Derived] Kern D, Ljotsson B, Lonndahl L, Hedman-Lagerlof E, Molander O, Liliequist B, Bradley M, Lindefors N, Kraepelien M. Self-Guided vs Clinician-Guided Online Cognitive Behavioral Therapy for Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2025 Feb 1;161(2):183-190. doi: 10.1001/jamadermatol.2024.5044. PMID 39693097
- [Derived] Kern D, Ljotsson B, Lonndahl L, Hedman-Lagerlof E, Bradley M, Lindefors N, Kraepelien M. Brief self-guided digital intervention versus a comprehensive therapist-guided online cognitive behavioural therapy for atopic dermatitis: a trial protocol for a randomised non-inferiority trial. BMJ Open. 2023 Feb 28;13(2):e068908. doi: 10.1136/bmjopen-2022-068908. PMID 36854583